CLINICAL TRIAL: NCT02688816
Title: Z 1313 - Comparison of Point-of-care Molecular Tests and Visual Inspection With Acetic Acid for Cervical Cancer Screening in HIV-infected Women in Lusaka, Zambia
Brief Title: Comparison of Cervical Cancer Screening Tests in HIV-infected Women in Lusaka, Zambia
Status: Completed | Type: Observational
Sponsor: Carla Chibwesha, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Carla Chibwesha, MD, Assistant Professor, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Other Study IDs: 14-0399; 3 D43 CA15378403S1 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2016-02-11; First posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Cervical Cancer
Keywords: visual inspection with acetic acid; Xpert HPV; OncoE6; screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women undergoing cervical cancer screening: HIV-infected women will undergo a cervical cancer screening examination using the VIA method. A digital photograph of the cervix will also be taken to aide visual screening. This is known as digital cervicography, and it is currently standard of care within cervical cancer screening clinics in Zambia.
  Cervical samples will be collected for molecular testing using Xpert HPV, and OncoE6. Cervical biopsy samples will also be obtained for confirmatory histopathologic diagnosis.
  Interventions: Device: Xpert HPV; Device: OncoE6

INTERVENTIONS:
Device: Xpert HPV — Point-of-care HPV DNA PCR test
Device: OncoE6 — Point-of-care E6 oncoprotein test

SUMMARY:
This study will compare the test performance characteristics of visual inspection with acetic acid (VIA), Xpert HPV, and OncoE6 in HIV-infected women, to inform the possible inclusion of these molecular tests in future cervical cancer screening

DETAILED DESCRIPTION:
This is a cross-sectional study taking place at cervical cancer prevention clinics in Lusaka, Zambia to determine the test performance characteristics (sensitivity, specificity, positive predictive value, and negative predictive value) of (1) visual inspection with acetic acid, (2) Xpert HPV, and (3) OncoE6 for the detection of CIN2+ among HIV-infected women. All cervical screening tests will be evaluated against a gold standard of histopathology obtained from cervical biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years and older.
* Women with documented HIV-infection in their medical record or by on-site testing through voluntary counseling and testing.
* Women willing to undergo pelvic examination and cervical cancer screening.
* Women willing to provide written, informed consent.

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected women undergoing cervical cancer screening in Lusaka, Zambia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Proportion of VIA-, Xpert HPV-, and OncoE6-positive results that are correctly identified | once, at the enrollment visit
  True positive rate (i.e., sensitivity) for CIN2+
Proportion of VIA-, Xpert HPV-, and OncoE6-negative results that are correctly identified | once, at the enrollment visit
  True negative rate (i.e., specificity) for CIN2+

CONTACTS AND LOCATIONS:
Overall Officials: Carla Chibwesha, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Adult Infectious Disease Centre at the University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson S, Dillner L, Elfgren K, Mints M, Persson M, Rylander E. A comparison of the human papillomavirus test and Papanicolaou smear as a second screening method for women with minor cytological abnormalities. Acta Obstet Gynecol Scand. 2005 Oct;84(10):996-1000. doi: 10.1111/j.0001-6349.2005.00702.x. PMID 16167918
- [Background] Abreu AL, Souza RP, Gimenes F, Consolaro ME. A review of methods for detect human Papillomavirus infection. Virol J. 2012 Nov 6;9:262. doi: 10.1186/1743-422X-9-262. PMID 23131123
- [Background] Bosch FX, Manos MM, Munoz N, Sherman M, Jansen AM, Peto J, Schiffman MH, Moreno V, Kurman R, Shah KV. Prevalence of human papillomavirus in cervical cancer: a worldwide perspective. International biological study on cervical cancer (IBSCC) Study Group. J Natl Cancer Inst. 1995 Jun 7;87(11):796-802. doi: 10.1093/jnci/87.11.796. PMID 7791229
- [Background] Davidson M, Schnitzer PG, Bulkow LR, Parkinson AJ, Schloss ML, Fitzgerald MA, Knight JA, Murphy CM, Kiviat NB, Toomey KE, et al. The prevalence of cervical infection with human papillomaviruses and cervical dysplasia in Alaska Native women. J Infect Dis. 1994 Apr;169(4):792-800. doi: 10.1093/infdis/169.4.792. PMID 8133094
- [Background] Elfgren K, Kalantari M, Moberger B, Hagmar B, Dillner J. A population-based five-year follow-up study of cervical human papillomavirus infection. Am J Obstet Gynecol. 2000 Sep;183(3):561-7. doi: 10.1067/mob.2000.106749. PMID 10992174
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Folpe AL, Agoff SN, Willis J, Weiss SW. Parachordoma is immunohistochemically and cytogenetically distinct from axial chordoma and extraskeletal myxoid chondrosarcoma. Am J Surg Pathol. 1999 Sep;23(9):1059-67. doi: 10.1097/00000478-199909000-00008. PMID 10478665
- [Background] Goel A, Gandhi G, Batra S, Bhambhani S, Zutshi V, Sachdeva P. Visual inspection of the cervix with acetic acid for cervical intraepithelial lesions. Int J Gynaecol Obstet. 2005 Jan;88(1):25-30. doi: 10.1016/j.ijgo.2004.09.018. PMID 15617701
- [Background] Gravitt PE, Paul P, Katki HA, Vendantham H, Ramakrishna G, Sudula M, Kalpana B, Ronnett BM, Vijayaraghavan K, Shah KV; CATCH Study Team. Effectiveness of VIA, Pap, and HPV DNA testing in a cervical cancer screening program in a peri-urban community in Andhra Pradesh, India. PLoS One. 2010 Oct 28;5(10):e13711. doi: 10.1371/journal.pone.0013711. PMID 21060889
- [Background] Grulich AE, van Leeuwen MT, Falster MO, Vajdic CM. Incidence of cancers in people with HIV/AIDS compared with immunosuppressed transplant recipients: a meta-analysis. Lancet. 2007 Jul 7;370(9581):59-67. doi: 10.1016/S0140-6736(07)61050-2. PMID 17617273
- [Background] Manos MM, Kinney WK, Hurley LB, Sherman ME, Shieh-Ngai J, Kurman RJ, Ransley JE, Fetterman BJ, Hartinger JS, McIntosh KM, Pawlick GF, Hiatt RA. Identifying women with cervical neoplasia: using human papillomavirus DNA testing for equivocal Papanicolaou results. JAMA. 1999 May 5;281(17):1605-10. doi: 10.1001/jama.281.17.1605. PMID 10235153
- [Background] Miller AB, Nazeer S, Fonn S, Brandup-Lukanow A, Rehman R, Cronje H, Sankaranarayanan R, Koroltchouk V, Syrjanen K, Singer A, Onsrud M. Report on consensus conference on cervical cancer screening and management. Int J Cancer. 2000 May 1;86(3):440-7. doi: 10.1002/(sici)1097-0215(20000501)86:33.0.co;2-a. No abstract available. PMID 10760836
- [Background] Mwanahamuntu MH, Sahasrabuddhe VV, Blevins M, Kapambwe S, Shepherd BE, Chibwesha C, Pfaendler KS, Mkumba G, Vwalika B, Hicks ML, Vermund SH, Stringer JS, Parham GP. Utilization of cervical cancer screening services and trends in screening positivity rates in a 'screen-and-treat' program integrated with HIV/AIDS care in Zambia. PLoS One. 2013 Sep 18;8(9):e74607. doi: 10.1371/journal.pone.0074607. eCollection 2013. PMID 24058599
- [Background] Mwanahamuntu MH, Sahasrabuddhe VV, Kapambwe S, Pfaendler KS, Chibwesha C, Mkumba G, Mudenda V, Hicks ML, Vermund SH, Stringer JS, Parham GP. Advancing cervical cancer prevention initiatives in resource-constrained settings: insights from the Cervical Cancer Prevention Program in Zambia. PLoS Med. 2011 May;8(5):e1001032. doi: 10.1371/journal.pmed.1001032. Epub 2011 May 17. PMID 21610859
- [Background] Mwanahamuntu MH, Sahasrabuddhe VV, Pfaendler KS, Mudenda V, Hicks ML, Vermund SH, Stringer JS, Parham GP. Implementation of 'see-and-treat' cervical cancer prevention services linked to HIV care in Zambia. AIDS. 2009 Mar 27;23(6):N1-5. doi: 10.1097/QAD.0b013e3283236e11. No abstract available. PMID 19279439
- [Background] Ngan HY, Garland SM, Bhatla N, Pagliusi SR, Chan KK, Cheung AN, Chu TY, Domingo EJ, Qiao YL, Park JS, Tay EH, Supakarapongkul W. Asia oceania guidelines for the implementation of programs for cervical cancer prevention and control. J Cancer Epidemiol. 2011;2011:794861. doi: 10.1155/2011/794861. Epub 2011 Apr 13. PMID 21559068
- [Background] Parkin DM. The global health burden of infection-associated cancers in the year 2002. Int J Cancer. 2006 Jun 15;118(12):3030-44. doi: 10.1002/ijc.21731. PMID 16404738
- [Background] Poljak M, Kocjan BJ. Commercially available assays for multiplex detection of alpha human papillomaviruses. Expert Rev Anti Infect Ther. 2010 Oct;8(10):1139-62. doi: 10.1586/eri.10.104. PMID 20954880
- [Background] Roden R, Wu TC. How will HPV vaccines affect cervical cancer? Nat Rev Cancer. 2006 Oct;6(10):753-63. doi: 10.1038/nrc1973. PMID 16990853
- [Background] Sankaranarayanan R, Nene BM, Shastri SS, Jayant K, Muwonge R, Budukh AM, Hingmire S, Malvi SG, Thorat R, Kothari A, Chinoy R, Kelkar R, Kane S, Desai S, Keskar VR, Rajeshwarkar R, Panse N, Dinshaw KA. HPV screening for cervical cancer in rural India. N Engl J Med. 2009 Apr 2;360(14):1385-94. doi: 10.1056/NEJMoa0808516. PMID 19339719
- [Background] Schiffman MH, Castle P. Epidemiologic studies of a necessary causal risk factor: human papillomavirus infection and cervical neoplasia. J Natl Cancer Inst. 2003 Mar 19;95(6):E2. doi: 10.1093/jnci/95.6.e2. No abstract available. PMID 12644550
- [Background] Schweizer J, Lu PS, Mahoney CW, Berard-Bergery M, Ho M, Ramasamy V, Silver JE, Bisht A, Labiad Y, Peck RB, Lim J, Jeronimo J, Howard R, Gravitt PE, Castle PE. Feasibility study of a human papillomavirus E6 oncoprotein test for diagnosis of cervical precancer and cancer. J Clin Microbiol. 2010 Dec;48(12):4646-8. doi: 10.1128/JCM.01315-10. Epub 2010 Oct 6. PMID 20926711
- [Background] Vedantham H, Silver MI, Kalpana B, Rekha C, Karuna BP, Vidyadhari K, Mrudula S, Ronnett BM, Vijayaraghavan K, Ramakrishna G, Sowjanya P, Laxmi S, Shah KV, Gravitt PE; CATCH Study Team. Determinants of VIA (Visual Inspection of the Cervix After Acetic Acid Application) positivity in cervical cancer screening of women in a peri-urban area in Andhra Pradesh, India. Cancer Epidemiol Biomarkers Prev. 2010 May;19(5):1373-80. doi: 10.1158/1055-9965.EPI-09-1282. PMID 20447927
- [Background] Zhao FH, Lewkowitz AK, Chen F, Lin MJ, Hu SY, Zhang X, Pan QJ, Ma JF, Niyazi M, Li CQ, Li SM, Smith JS, Belinson JL, Qiao YL, Castle PE. Pooled analysis of a self-sampling HPV DNA Test as a cervical cancer primary screening method. J Natl Cancer Inst. 2012 Feb 8;104(3):178-88. doi: 10.1093/jnci/djr532. Epub 2012 Jan 23. PMID 22271765
- See also: University of North Carolina website — http://www.unc.edu